CLINICAL TRIAL: NCT00136838
Title: Effect of Smoking Exposure on Tobacco Self-Administration Following Brief Abstinence
Brief Title: Effect of Smoking Exposure on Smoking Relapse Following Brief Abstinence - 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: #4725(2); R01DA017572 (NIH); R01DA017572-02 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco use
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neutral Cue first, then Active Cue (Experimental): Each participant receives two consecutive interventions.
  1. Neutral Cue: during this phase of treatment participants were presented with neutral (sham) cue
  2. Cigarette cue: during this phase of treatment participants were presented with active cigarette cue.
  Interventions: Behavioral: Neutral or active cigarette cues
- Active Cue first, then Neutral Cue (Experimental): Each participant receives two consecutive interventions.
  1. Cigarette cue: during this phase of treatment participants were presented with active cigarette cue.
  2. Neutral Cue: during this phase of treatment participants were presented with neutral (sham) cue
  Interventions: Behavioral: Neutral or active cigarette cues

INTERVENTIONS:
Behavioral: Neutral or active cigarette cues — Packets of cigarettes or cigarette smoke.

SUMMARY:
Recent research on the effects of nicotine on the brain and behavior presents an opportunity to advance medication development.

The purpose of this study is to develop a laboratory model for early-stage testing of new and existing treatments for nicotine addiction. Specifically, the investigators will develop a laboratory model of relapse to cigarette use in nicotine dependent volunteers.

DETAILED DESCRIPTION:
Tobacco use is the leading preventable cause of death in the United States. Recent research on the effects of nicotine on the brain and behavior presents an opportunity to advance medication development. The goal of this study is to develop a laboratory model for early-stage testing of new and existing compounds for the treatment of tobacco and nicotine addiction. In addition, the objective of this study is to develop a laboratory model of relapse induced by cigarette exposure that would reproduce the psychological and physiological processes that are involved when abstinent individuals progress from initial cigarette smoking (lapse) to a pre-abstinence level of use (relapse). Such a model may be used to study the mechanisms of relapse and to screen medications that might be effective in preventing relapse in treatment seekers.

This study will consist of two phases. Each phase will consist of a 5-day inpatient stay. During the first portion of inpatient stay, participants will not be permitted to smoke. During the second portion of inpatient stay, smoking reinstatement will be modeled, as participant will have opportunity to smoke, following the exposure to tobacco-related or control cues. A variety of behavioral, subjective, physiological, and performance measures will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nicotine dependence with psychological dependence
* Smokes at least 15 cigarettes per day for the three months prior to enrollment
* Currently not seeking treatment for nicotine dependence
* Medically healthy, on the basis of physical examination and medical history, vital signs, EKG, and laboratory tests
* Females must use an effective method of contraception for the duration of the study

Exclusion Criteria:

* Diagnosis of abuse or dependence on alcohol or drugs other than nicotine
* Current Axis I diagnosis or current treatment with psychotropic medications within the 3 months prior to enrollment
* History of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders
* Currently seeking treatment for nicotine disorders
* On parole or probation
* History of seizures or head trauma with loss of consciousness, brain contusion, or fracture
* History of significant recent violent behavior
* Blood pressure greater than 150/90
* History of eating disorders
* Pregnant

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2001-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve participants were recruited through advertisements in local newspapers and flyers.
Groups:
- Neutral Cue First, Then Active Cue: Participants receives two consecutive interventions in random order.
  1. Neutral Cue: during this phase of treatment participants were presented with neutral (sham) cue
  2. Cigarette cue: during this phase of treatment participants were presented with active cigarette cue
- Active Cue First, Then Neutral Cue: Each participant receives two consecutive interventions in random order.
  1. Cigarette cue: during this phase of treatment participants were presented with active cigarette cue
  2. Neutral Cue: during this phase of treatment participants were presented with neutral (sham) cue
Period: First Intervention ( 5 Days)
Arm/Group | Neutral Cue First, Then Active Cue | Active Cue First, Then Neutral Cue
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention ( 5 Days)
Arm/Group | Neutral Cue First, Then Active Cue | Active Cue First, Then Neutral Cue
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: This is a within-group study design, all participant who completed the study completed 2 phases of treatment, done in random order, each lasting 5 days and separated by at least 2 weeks. During one of the phases participants were exposed to active cigarette cues (pack of cigarettes, smoke) and during the other phase they were exposed to sham control cues (water bottle and the glass)
Arm/Group | Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Choice After 3 Day Abstinence
Description: Following 3 days of abstinence participants had an option to smoke cigarettes every 30 minutes for the maximum of 6 choices
Time Frame: During Day 4 experimental session
Measure: Mean (Standard Error); unit: number of cigarette choices (0-6)
Groups:
- Active Cue: During this phase participants were exposed to active cigarette cues: pack of cigarettes and a cigarette smoke
- Neutral Cue: During this phase of study participants were exposed to a neutral (sham) cue: a bottle of water and a glass
Arm/Group | Active Cue | Neutral Cue
Number analyzed (Participants) | 12 | 12
number of cigarette choices (0-6) | 2.50 (0.63) | 3.67 (0.58)

2. Other Pre Specified Outcome: Craving
Description: Measure of self-reported craving on a scale of 0-70 (0=no craving; 70= worst possible craving).
Time Frame: immediately following cue expose
Measure: Mean (Standard Error); unit: units on a scale (0-70)
Groups:
- Active Cue Craving; Neutral Cue Craving: intensity of craving following cue exposure
Arm/Group | Active Cue Craving | Neutral Cue Craving
Number analyzed (Participants) | 12 | 12
units on a scale (0-70) | 58.8 (3.1) | 53.8 (5.2)

ADVERSE EVENTS:
Time Frame: During the study
Groups:
- Neutral Cue: Neutral Cue: during this phase of treatment participants were presented with neutral (sham) cue
- Active Cue: 1.Cigarette cue: during this phase of treatment participants were presented with active cigarette cue.
Arm/Group | Neutral Cue | Active Cue
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes